CLINICAL TRIAL: NCT02428179
Title: StOP?-Trial: Impact of Structured Communication in the OR on Surgical Site Infections: Prospective Observational Clinical Trial
Brief Title: Impact of Structured Communication in the OR on Surgical Site Infections: Prospective Observational Clinical Trial
Acronym: StOP
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other); Triemli Hospital (Other); Kantonsspital Chur, Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: 161/14
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Incidence of Surgical Site Infection; Short Intraoperative Briefings; Mortality; Shared Mental Model
Keywords: Surgical site infection; Intraoperative briefings; Mortality; Wound closure; Surgical procedure
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group without Study intervention: Control group without Study intervention
  Interventions: Procedure: StOP? - Control group
- Group with Study intervention: Group with Study intervention
  Interventions: Procedure: StOP? - Intervention group

INTERVENTIONS:
Procedure: StOP? - Control group — Control group - Surgical procedure without Study Intervention
  Groups: Control group without Study intervention
Procedure: StOP? - Intervention group — Intervention group - Surgical procedure with intraoperative briefings, optional interventions: Transparent drape between anesthesia and sterile team, Controlling noise and potential distractors during wound closure, Nutritional support during the operation
  Groups: Group with Study intervention

SUMMARY:
Surgical site infection (SSI) is the most frequent complication in patients that undergo abdominal surgery. A previous prospective observational study in 167 patients undergoing elective open abdominal procedures showed that case-relevant communication protects from organ/space SSI whereas case-irrelevant communication during the last 20 minutes of the procedure is a risk factor for incisional SSI. Therefore, the introduction of a clinical applicable intervention "structured briefing using the StOP protocol" has been developed and was tested in pilot experiments. This intervention aims at improving case-relevant communication during the procedure and to reduce excess case-irrelevant communication at the end of an operation.

The hypothesis is: structured briefings during an operation reduce the incidence of SSI after surgery.

DETAILED DESCRIPTION:
Background

A number of publications has shown a relatively high rate of complications that are related to the treatment and not to the disease. Such iatrogenic incidents are an important influence on patient morbidity and increase healthcare costs. Therefore, patient safety and minimizing the risk of iatrogenic harm has become a major concern in healthcare. Surgical site infection (SSI) is one of the most frequent complication in patients that undergo surgery, leading to considerable costs.

In a previous study, the investigators established an empirical relationship between communication during surgery and SSI was shown in a prospective observational study in 167 patients undergoing major elective open abdominal procedures. An analysis of 11383 communication events observed by a team of trained work psychologists showed a relationship between intraoperative communication and SSI. Adjusted logistic regression analysis revealed that more case-relevant communication during the entire procedure was associated with a significant reduction in organ/space SSI (odds ratio 0.861, 95% confidence interval 0.750-0.987; P=0.034). Interestingly, case-irrelevant communication during the last 20 minutes of the procedure was associated with a significant increase of incisional SSI (odds ratio 1.1153, 95% confidence interval 1.040-1.196; P=0.002). Distractors such as noise and traffic were also assessed but had no effect on SSI. The current study is based on these observations, which reveal that case-relevant communication protects from organ/space SSI and case-irrelevant communication during the last 20 minutes of the procedure is a risk factor for SSI.

These findings can be interpreted in light of previous studies assessing communication in surgery and similar collaborative tasks which showed that explicit task-relevant communication fosters the development of a shared mental model of the task within the team. This facilitates coordination, because all team members are informed about the state of task progress, and can better anticipate their contribution. This is particularly important in critical phases of the procedure, as well as in OR teams composed of members with different levels of knowledge and expertise. Explicit task-related communication may be particularly useful to inform non-sterile team members (anesthetists, scrub nurses) that do not have full sight of the operative field at all times.

Although case-irrelevant communication in surgical teams has been found to foster a positive team-climate, it can be seen as a distractor if it diverts the attention away from the main task. This is more likely during the closing phase (last 20 minutes), because for most of the team members, the central task is already finished, and clearing and cleaning are routine tasks. If during routine tasks the team engages in too much non-patient relevant communication, attention to the closure may be diverted.

Given the previously found results, the introduction of a clinically applicable intervention (described below) has been tested in pilot studies. This intervention aims to assure a short discussion of case-relevant aspects at specific moments of the procedure, draw the attention of the on case-relevant communication during the main phase and to prevent a high increase in case-irrelevant communication at the end of an operation.

Objective

To perform a prospective clinical trial to test the impact of structured intraoperative briefings on SSI. The incidence of SSIs will be compared before and after the introduction of this intervention.

Methods

- Intraoperative briefings: First briefing: after exposure of the organ of interest, Second briefing: Intraoperative briefing before closure of the operative field.

* Trainings and Retrainings
* Optional Interventions: Transparent drape between anesthesia and sterile team; Controlling noise and potential distractors during wound closure; Nutritional support during the operation

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or emergency surgery

Exclusion Criteria

* Preexisting surgical site infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 3003 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical Site infections | 30 days postoperative

SECONDARY OUTCOMES:
Postoperative mortality | 30 days postoperative
Type of Operation / Laparoscopic procedure | 30 days postoperative
Grade of contamination | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Prof. Dr. med., Principal Investigator — Visceral and transplant surgery, University hospital, Berne
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

REFERENCES:
- [Result] Sax H, Uckay I, Balmelli C, Bernasconi E, Boubaker K, Muhlemann K, Ruef C, Troillet N, Widmer A, Zanetti G, Pittet D. Overall burden of healthcare-associated infections among surgical patients. Results of a national study. Ann Surg. 2011 Feb;253(2):365-70. doi: 10.1097/SLA.0b013e318202fda9. PMID 21217517
- [Result] Weber WP, Zwahlen M, Reck S, Feder-Mengus C, Misteli H, Rosenthal R, Brandenberger D, Oertli D, Widmer AF, Marti WR. Economic burden of surgical site infections at a European university hospital. Infect Control Hosp Epidemiol. 2008 Jul;29(7):623-9. doi: 10.1086/589331. PMID 18564917
- [Result] Mazzocco K, Petitti DB, Fong KT, Bonacum D, Brookey J, Graham S, Lasky RE, Sexton JB, Thomas EJ. Surgical team behaviors and patient outcomes. Am J Surg. 2009 May;197(5):678-85. doi: 10.1016/j.amjsurg.2008.03.002. Epub 2008 Sep 11. PMID 18789425
- [Result] Nurok M, Sundt TM 3rd, Frankel A. Teamwork and communication in the operating room: relationship to discrete outcomes and research challenges. Anesthesiol Clin. 2011 Mar;29(1):1-11. doi: 10.1016/j.anclin.2010.11.012. PMID 21295749
- [Result] Catchpole K, Mishra A, Handa A, McCulloch P. Teamwork and error in the operating room: analysis of skills and roles. Ann Surg. 2008 Apr;247(4):699-706. doi: 10.1097/SLA.0b013e3181642ec8. PMID 18362635